CLINICAL TRIAL: NCT03787979
Title: Effect of Increased Relative Stiffness of Lumbar Spine on Hamstrings Muscle Stretching in Individuals With History of Low Back Pain Suspected to Have a Clinical Lumbar Instability
Brief Title: Relative Stiffness of Lumbar Spine and Hamstrings Muscle Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Principal investigator, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/200.1010
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Back Pain; Instability Lumbar Spine; Muscle Tightness
Keywords: History of low back pain; Clinical lumbar instability; Stretching exercise
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either stretching exercise with lumbopelvic stiffening technique or lumbopelvic relaxing technique. They will be provided a 2-day wash-out period. Then, participants will cross-over to another technique.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor and investigator will be blinded to the random order. This process will be handled by the research manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbopelvic stiffening technique (Experimental): Hamstring muscle stretching with lumbopelvic stiffening technique.
  Interventions: Other: Lumbopelvic stiffening technique; Other: Lumbopelvic relaxing technique
- Lumbopelvic relaxing technique (Active Comparator): Hamstrings muscle stretching with lumbopelvic relaxing technique.
  Interventions: Other: Lumbopelvic stiffening technique; Other: Lumbopelvic relaxing technique

INTERVENTIONS:
Other: Lumbopelvic stiffening technique — Participants will stretch their hamstrings muscle in standing position with lumbopelvic stiffening technique. Fifteen percent of the body weight will be used to standardize stretching force. During stretching protocol, the participants will be instructed to face the hydraulic table with their hips square, maintain trunk straight up and look straight ahead. Researcher commands "during adjusting the bed up, please tense your back rigid". After that, hydraulic bed will be lifted up until force reaches 15 percent of the body weight. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions.
Other: Lumbopelvic relaxing technique — Participants will be instructed to face the hydraulic table with their hips square, maintain trunk straight up and look straight ahead. The researcher commands "During adjusting the bed up, please relax your back". The hydraulic bed will be lifted up until force reaches 15 percent of the body weight. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions.

SUMMARY:
The purpose of this study is to investigate the effect of lumbopelvic stabilization on hamstrings muscle stretching in individuals with history of low back pain suspected to have a clinical lumbar instability.

DETAILED DESCRIPTION:
The participants between the age of 20 and 40 years with history of low back pain will be recruited from Mahidol University using a poster posted at Faculty of Physical Therapy. All participants will be explained the purposes, advantages, disadvantages and procedures of the study by the researcher. The participant will be asked to sign an informed consent if the participants are willing to participate in this study.

After obtaining the written informed consent, the researcher, who works in musculoskeletal system including low back pain for 7 years and has received 3 training sessions on clinical observation of aberrant movement, will perform 2 clinical tests including clinical observation of aberrant movement patterns and passive straight leg raising test to identify clinical lumbar instability, and measure hamstrings muscle length using clinical motion analysis system. The researcher will also screen for exclusion criteria using a check list.

For those who are qualified for the study, the participants will be asked to fill out the demographic data and physical activity questionnaire. The researcher will perform additional clinical examination including modified Thomas test, back extensor muscle strength test assessed by a handheld dynamometer, Trendelenburg's test and lumbar stability test. After clinical tests, lumbopelvic, pelvic, and lumbar range of motions during an active forward bend task will be measured by using the clinical motion analysis system. These outcome measures will be assessed for baseline (Pre-1). After baseline data collection, the participants will be divided into 2 groups; lumbopelvic stiffening group (LS) or lumbopelvic relaxing group (LR) by randomly generated code in a concealed envelope.

The participants in LS group will stretch the hamstrings muscle in standing position with lumbopelvic stabilization. Fifteen percent of the body weight will be used to standardize stretching force. This force will be controlled by visual feedback from load cell. During stretching protocol, the participants will be instructed to face the hydraulic table with the hips square, maintain trunk straight up and look straight ahead. Researcher commands "during adjusting the bed up, please tense the lower back rigid". After that, hydraulic bed will be lifted up until force reaches 15 percent of the body weight. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions. To ensure that participant correctly performs lumbopelvic stabilization, the researcher will palpate at ASIS and iliac crest to check pelvic motion during hamstrings muscle stretching. Pelvic motion indicates loss of lumbopelvic stabilization. Participant will be asked to re-perform another repetition. Our protocol is based on a previous study by DePino et al., 2000. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions. The investigators use 30 seconds because a systematic review suggests that 30 seconds is the most effective dose for hamstrings muscle stretching.

For the participants in LR group, the participants will be instructed to face the hydraulic table with the hips square, maintain trunk straight up and look straight ahead. The researcher commands "During adjusting the bed up, please relax the lower back". The hydraulic bed will be lifted up until force reaches 15 percent of the body weight. Participant will perform 30 seconds/repetition for 4 repetitions with 15 seconds rest between repetitions.

After the intervention, the participants will be reassessed for hamstrings muscle length test, lumbar motion, pelvic motion and total lumbopelvic motion (Post-1). Because this study uses a cross-over study design, participants will be asked to maintain the usual physical activity for 2 days as a wash-out period. Then, the participants will be re-assessed for baseline data (Pre-2), and cross-over to another stretching group (LS changes to LR, while LR changes to LS). After completion of intervention, the participants will be re-assessed for post-intervention (Post-2). These to determine the effectiveness of lumbopelvic stabilization during hamstrings stretching in standing.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 20 and 40
2. A recurrent pattern of LBP at least two episodes that interfered with activities of daily living and/or required treatment
3. Presenting aberrant movement pattern during active forward bend test
4. Passive straight leg raising test (SLR) greater than 91 degrees
5. Having hamstrings muscle tightness of both legs (passive knee extension in supine with 90° hip flexion position greater than 20 degrees)

Exclusion Criteria:

1. Having a history of abdominal, back surgery and/or fracture.
2. Having any red flags, such as infection, tumor, fracture, radicular syndrome, or inflammatory.
3. Pregnancy or having menstruation.
4. Having spinal deformities, such as scoliosis.
5. Having neurological, musculoskeletal or cardiopulmonary diseases.
6. Previously receiving physical therapy intervention involving in motor control training.
7. Taking muscle relaxant medication.
8. Having hip joint stiffness or pain
9. Having positive Trendelenburg's sign.
10. Currently having routine vigorous exercise.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Lumbar, pelvic, and lumbopelvic motions at baseline. | These data will be collected at baseline and immediately after intervention.
  Clinical motion analysis system will be used to measure these segmental motions. This system is composed of triple axis accelerometers (MPU6050, China), data acquisition board (Arduino Uno R3, Italy), and a LabVIEW software version 2012 (National Instrument, USA). The system will be used to measure pre- and post-intervention of angle of lumbar, pelvic, and lumbopelvic motions through a custom LabVIEW program at 100 Hz.
Lumbar, pelvic, and lumbopelvic motions after intervention. | These data will be collected at immediately after intervention.
  Clinical motion analysis system will be used to measure these segmental motions. This system is composed of triple axis accelerometers (MPU6050, China), data acquisition board (Arduino Uno R3, Italy), and a LabVIEW software version 2012 (National Instrument, USA). The system will be used to measure pre- and post-intervention of angle of lumbar, pelvic, and lumbopelvic motions through a custom LabVIEW program at 100 Hz.
Hamstrings muscle length at baseline. | These data will be collected at baseline.
  Clinical motion analysis system will be used to measure the angle of knee extension that represents hamstrings muscle length at pre- and post-intervention.
Hamstrings muscle length after intervention. | These data will be collected at immediately after intervention.
  Clinical motion analysis system will be used to measure the angle of knee extension that represents hamstrings muscle length at pre- and post-intervention.

SECONDARY OUTCOMES:
Muscle length based on modified Thomas and Trendelenburg test. | These data will be collected at baseline only.
  Clinical tests will be performed at the baseline because they could be a potential confounding factor.
Abdominal and back muscle strength . | These data will be collected at baseline only.
  Abdominal and back muscle strengths will be measured by using a hand-held dynamometer. Clinical tests will be performed at the baseline because they could be a potential confounding factor.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The IPD of this study will be shared upon official request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The supporting information will be sent upon official request.
Access Criteria: Having an official written request.

REFERENCES:
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Sahrmann S, Azevedo DC, Dillen LV. Diagnosis and treatment of movement system impairment syndromes. Braz J Phys Ther. 2017 Nov-Dec;21(6):391-399. doi: 10.1016/j.bjpt.2017.08.001. Epub 2017 Sep 27. PMID 29097026
- [Background] Jandre Reis FJ, Macedo AR. Influence of Hamstring Tightness in Pelvic, Lumbar and Trunk Range of Motion in Low Back Pain and Asymptomatic Volunteers during Forward Bending. Asian Spine J. 2015 Aug;9(4):535-40. doi: 10.4184/asj.2015.9.4.535. Epub 2015 Jul 28. PMID 26240711
- [Derived] Wattananon P, Prasertkul W, Sakulsriprasert P, Laskin JJ. Effect of increased relative stiffness of the lumbar spine on hamstring muscle stretching in individuals with a history of low back pain suspected to have a clinical lumbar instability: A randomized crossover design. Clin Biomech (Bristol). 2020 May;75:104996. doi: 10.1016/j.clinbiomech.2020.104996. Epub 2020 Apr 20. PMID 32339943